CLINICAL TRIAL: NCT05359367
Title: A Novel Approach to the Development of New Treatment Strategies to Enhance True Recovery After Stroke, Based on Laboratory Movement Analysis and Clinical Aspects of Gait Function and Walking
Brief Title: A Novel Approach to Enhance True Recovery After Stroke
Status: Terminated | Type: Observational
Why Stopped: Due to low recruitment and follow up rate.
Sponsor: Danderyd Hospital (Other)
Collaborators: KTH Royal Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-05430-01
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Inpatients; Recovery of Function; Observational Study
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Observational — Laboratory movement analysis, navigated transcranial magnetic stimulation and clinical aspects of gait function and walking.

SUMMARY:
The purpose of this study is to elucidate pathophysiological mechanisms behind gait disturbances during the early recovery phase after hemiparetic stroke to identify targets for new treatment strategies.

Using an explorative, observational study design, pathophysiological mechanisms at play during the early recovery phase will be monitored, by repeated clinical assessments during inpatient rehabilitation as well as examinations of muscle activation patterns, kinematics of walking, corticospinal and reticulospinal function < 1 month, 3 and 6 months after hemiparetic stroke.

Inclusion: Eligible patients will have suffered a stroke, verified by CT or MRI examination and are admitted to inpatient care at the University Department of Rehabilitation Medicine Danderyd Hospital (RUDS). Thirty patients will be included consecutively. With an anticipated loss of 4-10 patients, at least 20 are expected to complete the study.

The clinical assessment protocols include standardized measures for the assessment of clinical and self-perceived aspects of functioning and disability. These assessments will be performed and repeated < 1 month, at 3 months and 6 months post-stroke by a therapist not responsible for rehabilitation interventions. At each of these assessment instances, laboratory movement analysis including electromyography (EMG) and ultrasound of the lower extremity muscle will be performed. In addition, a short assessment of body function and activity will be performed weekly during inpatient rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Participants with hemiplegia, dependence in ambulation (1- 4 according to the Functional Ambulation Categories (FAC)),
* >= 50 points on the Trunk Control Test.
* Impaired dorsiflexion manifested as impaired voluntarily dorsiflexion and inability to hold the ankle in a dorsiflexed position while sitting, and for ambulatory participants, impaired dorsiflexion during swing phase and initial contact during visual inspection of gait.
* Recommended for an ancle foot orthosis (AFO) by an experienced physiotherapist. Able to understand study information and provide informed consent.

Exclusion Criteria:

* Contracture that severely restricts gait movements in a lower limb joint,
* cardiovascular or other somatic condition incompatible with intensive gait training,
* notifiable infectious disease, contagious infections (e.g. MRSA or ESBL)
* Inability to participate in the rehabilitation intervention due to behavioral or psychiatric disorder
* when magnetic resonance imaging will be performed, additional exclusion criteria are current or history of epilepsy, metal implants in the brain/skull cochlear implants, any implanted neurostimulator, cardiac pacemaker or cardiac implants of metal and infusion device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will have suffered a stroke, verified by CT or MRI examination and are admitted to inpatient care at the University Department of Rehabilitation Medicine Danderyd Hospital.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer score (FMA-LE) | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Assesses sensory and movement related functions in the lower extremity (0p max impairment summed up to 86p max no detected impairment)

SECONDARY OUTCOMES:
Motion analysis during gait | At baseline, at 3 and 6 months to assess change.
  In a movement laboratory (Vicon V16), data for motion analysis will be collected by assessing orientation of body segments and joint angle trajectories and forces by means of force plates (AMTI) during walking.
Electromyography (EMG) | At baseline, at 3 and 6 months to assess change.
  EMG is used to measure muscle activation patterns during gait.
Neuroflexor | At baseline, at 3 and 6 months to assess change.
  Medical technology device. Assesses spasticity by identifying the neural, viscous and elastic components during passive movement using a biomechanical algorithm (presented in Newton)
Modified Ashworth scale 0-5 | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Assesses spasticity on a 6 point scale/muscle (0p no impairment, 5p max impairment/muscle)
Passive range of motion in the lower extremity | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Clinical assessment of range of motion with a goniometer
The 10 meter walk test | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Assesses gait speed
6 minutes walk test | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Assesses walking endurance in meters walked
Rated Perceived Exertion (RPE) Scale | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Ratings (min 6, max 20) according to the RPE scale are made at the end of the 6 minutes walk test.
The Functional Ambulation Categories (FAC) | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Assesses independence in walking (0p nonfunctional, 5p independent) Total score 0-5p
The Balance evaluation systems test (BEST-test) | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Assesses postural control, incorporating bio-mechanical systems, limits of stability, anticipatory postural adjustment, automatic postural responses, sensory orientation, stability in gait (0p max impairment summed up to 108p no impairment)
Falls Efficacy Scale (FES-S) | At baseline and at 3 and 6 months to assess change.
  Assesses self perceived balance in every day life activities rated on a 11 point scale (0p not safe at all 10p completely safe). Total score: 0- 130 p
Navigated Transcranial magnetic stimulation (nTMS) | At baseline and at 3 and 6 months to assess change.
  To estimate the integrity of the corticospinal tract, transcraniel magnetic stimulation will be applied to the primary motor cortex and motor evoked potentials will be will be recorded from the lower leg muscles using electromyography.
The Montreal Cognitive Assessment (MoCa) | At baseline and at 3 and 6 months to assess change.
  Assesses mental function (0p max impairment summed up to 30p no detected impairment)
National Institute of Health Stroke Scale | At baseline and at 3 and 6 months to assess change.
  To assess overall effects of stroke (ranging from 0-44 points, a higher score indicating more severe disability).
Barthel Index | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Assesses independence in mobility and personal care (0p dependent 10/15p independent) Total score 0-100p
Monofilament | At baseline, at 3 and 6 months to assess change.
  Measuring cutaneous sensory perception threshold under foot with a pressure of 4, 6 and 10 grams.
Pain drawing | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Self-assessed location and type of pain on the body
Numeric rating scale of pain | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Self-rated general intensity of pain at time of assessment (0 no pain, 10 worst imaginable pain)
Medical Research Council scale | At baseline, weekly during inpatient rehab and at 3 and 6 months to assess change.
  Assesses movement strength at a specific joint and motion (0 no muscle activity 5 normal force)
Walking impact scale (Walk-12) | At baseline and at 3 and 6 months to assess change
  Measures rated limitations in walking activities (1 no limitation, 5 extreme limitation)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Palmcrantz, PhD, Principal Investigator — Dep of Clinical Sciences, Karolinska Institutet
Locations (1):
- Department of Rehabilitation Medicine, Danderyd Hospital, Danderyd, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No